CLINICAL TRIAL: NCT04994626
Title: Phase II, Multi-Center Study to Evaluate the Efficacy and Safety of Ibrutinib Combined With Rituximab for Treatment of Relapsed Refractory MYD88 and CD79A/B (or CD79B Alone) DLBCL Who Have Received at Least Two Prior Therapies
Brief Title: Ibrutinib Combined With Rituximab for Treatment of Relapsed Refractory MYD88 and CD79A/B (or CD79B Alone) DLBCL Who Have Received at Least Two Prior Therapies
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2613
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: DLBCL; MYD88 Gene Mutation; CD79A Gene Mutation; CD79B Gene Mutation; Relapse; Refractory Lymphoma
Keywords: R/R DLBCL; MYD88 Gene Mutation; CD79A/B Gene Mutation; Ibrutinib; Rituximab
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibrutinib Combined With Rituximab (Experimental): Induction therapy: Ibrutinib 560mg administered oral once a day of each 21-day cycle for 6 cycles. Rituximab 375mg/m² administered intravenously (IV) on Day 1 of each 21-day cycle for 6 cycles.
  Maintenance therapy: Ibrutinib 560mg administered oral once a day of each 56-day cycle for 6 cycles. Rituximab 375mg/m² administered intravenously (IV) on Day 1 of each 56-day cycle for 6 cycles.
  Interventions: Drug: Ibrutinib Combined With Rituximab

INTERVENTIONS:
Drug: Ibrutinib Combined With Rituximab — Drug: ibrutinib ibrutinib 560mg administered orally once daily. Other Name: Imbruvica
  Drug: rituximab rituximab 375mg/m² administered intravenously (IV)
  Other Names: Imbruvica Combined With Rituximab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ibrutinib Combined With Rituximab in Relapsed Refractory MYD88 and CD79A/B (or CD79B Alone) DLBCL Who Have Received at Least Two Prior Therapies.

DETAILED DESCRIPTION:
Recent studies have found that about 30% of DLBCL have mutations in MYD88 and/or CD79A/B genes. MYD88 and CD79A/B protein molecules belong to two signal transduction pathways, which regulate B cell proliferation. Both MYD88 and CD79A/B gene mutations can abnormally activate BTK located downstream of MYD88 and CD79A/B, leading to over activation and proliferation of B cells.

Ibrutinib is the first generation of oral BTKi, which may theoretically inhibit the tumorigenesis of DLBCL with abnormal BTK activation caused by mutations in MYD88 and CD79A/B genes.

A phase II clinical study of ibrutinib monotherapy in the treatment of relapsed and refractory DLBCL showed that the effective rate of ibutinib for single CD79B mutation was 55.5% (5/9 cases), and that for both CD79B and MYD88 mutations was 80% (4/5 cases). About 40 ~ 50% of primary central nervous system large B cell lymphoma (PCNSL) have CD79B and MYD88 mutations. A small sample study found that the overall response rate (ORR) for the treatment of relapsed and refractory PCNSL with ibrutinib was 77% (10/13). An expanded sample study of 44 cases of PCNSL treated with ibrutinib found that the ORR is 52% and progression-free survival (PFS) is 4.8 months. These results suggest that ibrutinib may be more effective in DLBCL with MYD88 and CD79A/B or CD79B mutations.

The relationship between mutations in MYD88 and CD79B and therapeutic sensitivity of ibrutinib can not be simply categorized, because abnormalities in other genes of B cell signaling pathway, such as CARD11, TNFAIP3, CXCR4, JAK1 and PIM1, may also affect the efficacy of ibrutinib. Therefore, it is necessary to comprehensively analyze the gene abnormalities of other B cell related signaling pathways, such as downstream signal of Bruton kinase, CXCR, JAK-STAT, and NFKB, to find out the most effective group of DLBCL patients treated with ibrutinib.

This phase II, single-arm, open-label, multi-center clinical trial will evaluate the efficacy and safety of ibrutinib combined with rituximab in treating relapsed refractory MYD88 and CD79A/B (or CD79B alone) DLBCL who have received at least two prior therapies. The study will also explore the relationship between MYD88 and/or CD79A/B and efficacy, and detect the gene abnormality by Next Generation Sequencing (NGS) and evaluate the relationship between other gene abnormality and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to understand and be willing to sign a written informed consent document;
2. Men and woman who are at least 18 years of age on the day of consenting to the study;
3. According to the WHO 2016 classification criteria, pathologically confirmed CD20+diffuse large B-cell lymphoma;
4. Patients with MYD88 and CD79A/B mutations or CD79B alone;
5. Relapse or progression after treatment with at least two prior therapies;
6. There is at least one measurable lesion, defined as a two-path measurable, intraductal lesion short neck >1.5cm, extranodal lesion short diameter >1.0cm;
7. Eastern Cooperative Oncology Group (ECOG) performance status =< 2
8. Blood routine examination meets the following criteria:

   Neutrophil count ≥ 1.0 x 109 / L; Platelet ≥ 75 x 109 / L; Hemoglobin ≥ 10.0 g / dL;
9. The main organ function meets the following criteria:

   Aspartate aminotransferase and alanine aminotransferase ≤ 2.0 times the upper limit of normal value; Bilirubin ≤ 2.0 mg / dL; Creatinine clearance rate ≥ 60 mL / min;
10. Must agree to effective contraception

Exclusion Criteria:

1. Transformed diffuse large B-cell lymphoma;
2. HBV DNA positive or HCV RNA positive;
3. Patient is known to have an uncontrolled active systemic infection;
4. Left ventricular ejection fraction < 40%;
5. Previous autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, dry syndrome, ankylosing spondylitis, etc;
6. Immunosuppressive drugs are being or have been used in the past;
7. Known hypersensitivity to the study drug or any of its excipients;
8. There are other active malignant tumors that may interfere with this study requiring treatment;
9. Known history of human immunodeficiency virus (HIV) infection;
10. Previous autologous stem cell transplantation or allogeneic hematopoietic stem cell transplantation;
11. The investigator judges that the patient has other inappropriate circumstances.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | 24 months after the last patient's enrollment
  The ORR includes complete response and partial response. The treatment response assessments are as follows: Evaluation of treatment response are performed every 2 cycles followed the International Lymphoma Collaborative Group guidelines.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | at 6 month and 1 year
  From the date into this study to disease progression or death
Overall Survival (OS) | at 6 month and 1 year
  From the date into this study to death
Event Free Survival (EFS) | at 6 month and 1 year
  From the date into this study to disease progression, relapse from CR as assessed by the investigator, completion of study treatment followed by subsequent systemic anti-lymphoma therapy, or death from any cause, whichever occurred first.
Adverse events | 24 months after the last patient's enrollment
  AEs will be evaluated using the NCI CTCAE v4.0.
Assessment of the correlation between MYD88 and/or CD79A/B or other gene abnormality and efficacy. | 24 months after the last patient's enrollment
  To explore the relationship between MYD88 and/or CD79A/B and efficacy and to detect the gene abnormality by Next Generation Sequencing (NGS) and evaluate the relationship between other gene abnormality and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D., Principal Investigator — Cancer Hospital Chinese Academy of Medical Sciences & Peking Union Medical College

IPD SHARING:
Plan to Share IPD: No